CLINICAL TRIAL: NCT02777489
Title: Influence of Single Nucleotide Polymorphisms of Carboxypeptidase D (CPD) Gene on Body Weight and Fat Mass Reduction by Perindopril in Obese Subjects: A Phase II, Multicenter, Double-blind Study
Brief Title: Influence of Carboxypeptidase D (CPD) Gene on Body Weight and Fat Mass Reduction by Perindopril in Obese Subjects
Acronym: GPD-01-01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unproven hypothesis
Sponsor: Gene PreDiT (Industry)
Collaborators: Blueclinical, Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GPD-01-01
Record Dates: First submitted 2016-03-07; First posted 2016-05-19 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Obesity
Keywords: obesity; perindopril; carboxypeptidase D; genotyping; theranostic
MeSH Terms: conditions — Obesity | interventions — Perindopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perindopril Bluepharma 8 mg (Experimental): Each participant will have an at least 4-week run-in period, followed by a 6 weeks treatment period with Perindopril 8 mg.
  Interventions: Drug: Perindopril

INTERVENTIONS:
Drug: Perindopril — Perindopril Bluepharma 8 mg tablets, daily, during approximately 12 weeks

SUMMARY:
The primary objective of this study is to evaluate the Carboxipeptidase D (CPD) genotyping as a predictive biomarker of body weight and/or fat mass reduction in obese patients treated with perindopril.

There is nonclinical and clinical evidence that a subgroup of human subjects may present a decrease in body weight and/or fat mass following treatment with perindopril. Although the individual characteristics that determine such effect are still unknown, Gene PreDiT SA (Biocant Park, Cantanhede, Portugal) discovered that certain genetic characteristics (e.g., single nucleotide polymorphisms (SNPs) of CPD gene) may play a role and potentially could serve as a potential predictive biomarker of response to perindopril.

These promising results, along with the fact that perindopril is a medicine already in use in clinical practice, led Gene PreDiT SA to decide to proceed with the development of a theranostic approach for the treatment of obesity. Such theranostic approach consists on the use of CPD genotyping to identify obese subjects that could present improved body weight and fat mass reduction following treatment with perindopril.

The current clinical trial aims to prove the concept and provide data to design further confirmatory studies. Additionally this study will evaluate the association between CPD SNPs genotypes and response to perindopril; the effect of perindopril in waist circumference, waist/hip ratio, and BMI and the tolerability and safety of perindopril in the study population.

DETAILED DESCRIPTION:
The study consists of 2 periods and 4 visits (V): a run-in period of at least 4 weeks (V1 to V2) and a 12-week perindopril treatment period (V2 to V4).

After written informed consent, patients will undergo screening evaluations (V1). Patients who meet the selection criteria will enter a run-in period of 4 weeks where they will be given dietary and exercise counseling as standardized non-drug therapy. After the run-in period (V2), patients will start the pharmacological therapy period where they will receive perindopril 8 mg, once daily, for 12 weeks, concomitantly with the previously established standardized non-drug therapy.

During the 12-week pharmacological treatment, patients will attend an intermediate study visit (V3) at approximately 6 weeks and a final visit (V4) for efficacy and safety assessments.

Body weight, body mass index (BMI), waist and hip circumference, and body fat mass estimation will be assessed at every study visit.

A total of 160 subjects will be enrolled, to have approximately 120 subjects evaluable.

After V2, patients will be administered perindopril 8 mg, once daily, for 12 weeks, concomitantly with the previously established standardized non-pharmacological therapy.

Blood sampling for clinical safety laboratory assessments (hematology and plasma biochemistry) will be collected at the screening, at the end of the run-in period, at the intermediate treatment visit, and at the end of the perindopril treatment period.

At the screening, blood will also be collected for CPD genotyping, but the results will remain blinded until database closure.

Safety will be evaluated through the assessment of treatment-emergent adverse events, vital signs and clinical laboratory tests. Adverse events will be monitored throughout the study. Vital signs will be recorded at each scheduled visit. Clinical safety laboratory parameters will be collected at screening, end of the run-in period, at the intermediate treatment visit, and at the end of the treatment period.

Abnormalities in vital signs and laboratory parameters will be assessed by the clinical investigator in terms of clinical relevance. Clinically significant abnormalities in clinical laboratory and vital signs will be reported as adverse events.

Associations between CPD SNPs genotypes and patient response will be assessed through the appropriate statistical methods. The primary efficacy analysis will compare the response rate in the group of subjects with the SNPs of interest and the group of the remaining subjects. A logistic regression model will be used to assess the group differences. Weight and fat mass at the start of the perindopril treatment period and gender will be used as covariates. Other covariates will be investigated for exploratory purposes, but will not be included in the model where main treatment effects are tested and compared. All the secondary efficacy endpoints will be assessed using analysis of covariance (ANCOVA). In general, the principles applied for the primary efficacy analysis will be replicated for the secondary efficacy analysis.

Adverse events will be tabulated and summarized according to system organ class (SOC) and preferred term (PT).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Man or woman with 18 years or more;
* Body Mass Index (BMI) between 30.0 to 40.0 kg/m2;
* Willingness and ability to comply with the study requirements;
* Ability to understand and sign informed consent;
* If woman of childbearing potential, she agrees to adopt effective contraceptive methods.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* History of obesity with a known cause (e.g., hypothyroidism, Cushing's disease);
* Under treatment with perindopril or other angiotensin converting enzyme (ACE) inhibitor, or with an angiotensin receptor blocker (ARB) or a renin inhibitor;
* Hypertension diagnosed at screening;
* Significant variation in weight (more 10%) in the past 3 months before screening visit;
* History of anorexia nervosa, bulimia, or binge-eating disorder;
* Systolic blood pressure <110 mmHg;
* History of hypersensitivity to perindopril, or related compounds, or to any of the inactive ingredients;
* History of angioedema associated with previous ACE inhibitor therapy;
* History of idiopathic or hereditary angioedema;
* Treatment with concomitant medication affecting weight loss (e.g. metformin) starting within the 3 months prior to screening;
* Treatment with concomitant medication that might interfere with the absorption, distribution, metabolism or elimination of perindopril, or, is likely to compromise the safety of subject (e.g. diuretics in patients with salt and/or volume depletion, insulin or oral antidiabetics in patients prone to develop hypoglycemic episodes, lithium, vasodilators in patients prone to develop hypotension, tricyclic antidepressants, antipsychotics, anesthetics, gold, potassium supplements or potassium-containing salt substitutes);
* Treatment with any investigational drug or device within 1 month before the start of the run-in period;
* Moderate to severe hepatic impairment (Child-Pugh score ≥ 7) or moderate to severe renal impairment (glomerular filtration rate (GFR) ≤ 59 ml/min);
* Unstable coronary artery disease;
* Aortic and mitral valve stenosis / hypertrophic cardiomyopathy
* Hemodialysis patients;
* Kidney transplantation;
* Anaphylactoid reactions during low-density lipoproteins (LDL) apheresis;
* Neutropenia/agranulocytosis/thrombocytopenia/anemia;
* Patients undergoing major surgery or during anesthesia with agents that produce hypotension;
* Hyperkalemia;
* Any other condition or therapy that the study physician considers to make the subject unsuitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-02-18; Primary Completion 2017-01-18 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Response rate, defined as the proportion of patients who will lose at least 3% of body weight and/or at least 3% of fat mass from end of the run-in period to the end of the perindopril treatment period. | From end of the run-in period to the end of the perindopril treatment period, up to 12 weeks

SECONDARY OUTCOMES:
End vs start of treatment relative change in body weight. | From end of the run-in period to the end of the perindopril treatment period, up to 12 weeks
End vs start of treatment relative change in fat mass. | From end of the run-in period to the end of the perindopril treatment period, up to 12 weeks
End vs start of treatment relative change in waist circumference. | From end of the run-in period to the end of the perindopril treatment period, up to 12 weeks
End vs start of treatment relative change in hip circumference. | From end of the run-in period to the end of the perindopril treatment period, up to 12 weeks
End vs start of treatment relative change in fasting lipid profile. | From end of the run-in period to the end of the perindopril treatment period, up to 12 weeks
Frequency and type of adverse events. | From V1 until the end of the perindopril treatment period, , up to 16 weeks
Response rate, defined as the proportion of patients who will lose at least 5% of body weight and/or at least 5% of fat mass from end of the run-in period to the end of the perindopril treatment period. | From end of the run-in period to the end of the perindopril treatment period, up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (13):
- Portugal (13):
  - Unidade de Saúde Familiar Escariz, Arouca
  - Centro Hospitalar do Baixo Vouga (CHBV), EPE, Aveiro
  - Unidade de Saúde Familiar Canelas, Canelas
  - Centro Hospitalar Cova da Beira (CHCB), EPE, Covilha
  - Unidade de Saúde Familiar Lethes, Ponte de Lima
  - Centro Hospitalar de São João (CHSJ), E.P.E, Porto
  - Unidade de Saúde Familiar Arca d'Água, Porto
  - Unidade de Cuidados de Saúde Personalizados Carvalhido, Porto
  - Unidade Local de Saúde do Alto Minho (ULSAM), E.P.E., Viana do Castelo
  - Unidade de Saúde Familiar Nova Salus, Vila Nova de Gaia
  - Unidade de Saúde Familiar Santo André de Canidelo, Vila Nova de Gaia
  - Centro Hospitalar V.N.Gaia/Espinho (CHVNG/E)- Endocrinology, Vila Nova de Gaia
  - Centro Hospitalar Vila Nova de Gaia/Espinho (CHVNG/E), Vila Nova de Gaia